CLINICAL TRIAL: NCT04216771
Title: Randomized Comparison of Consolidation Treatment in Elderly Patients With Acute Myeloid Leukemia: Idarubicin (IDA) Combined With Intermediate-dose Cytarabine Versus Intermediate-dose Cytarabine Alone
Brief Title: Comparing the Consolidation Regimens of IDA With Intermediate-dose Cytarabine Versus Intermediate-dose Cytarabine Alone for Elderly AML Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Jianda Hu, Director of the department of Hematology, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AML-19-01
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: AML in Remission
MeSH Terms: interventions — Idarubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IDA with ID Cytarabine (Experimental)
  Interventions: Drug: Idarubicin; Drug: ID cytarabine
- ID Cytarabine (Active Comparator)
  Interventions: Drug: ID cytarabine

INTERVENTIONS:
Drug: Idarubicin — Idarubicin 10mg/m²/day, D1 (IV)
  Arms: IDA with ID Cytarabine
Drug: ID cytarabine — Cytarabine 1.5g/m² /12h, D1-D3 (IV)

SUMMARY:
This study evaluates Idarubicin (IDA) in combination with the intermediate-dose cytarabine, compared with intermediate-dose cytarabine alone, as a consolidation treatment for elderly AML in first remission.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed de novo AML who achieved complete remission (CR), including CRi and CRp after a maximum number of 2 cycles of induction chemotherapy.
* Histologically or morphologically confirmed diagnosis of AML except for AML M3 (acute promyelocytic leukemia)
* No contraindication to anthracyclines : decompensated or uncontrolled heart failure, recent myocardial infarction, current signs of cardiac impairment, uncontrolled arrhythmias, LVEF (left ventricular ejection fraction) < 50%
* Age ≥ 60 years and < 75 years
* ECOG performance status ≤2
* Written informed consent
* No psychological, familial, social, or geographic reason that would compromise clinical follow up

Exclusion Criteria:

* Relapsed or refractory AML
* Patients with acute promyelocytic leukemia (APL)
* Patients with secondary type AML (post myelodysplastic syndrome MDS or therapy-related AML)
* Severe pshyciatric or organic disorder, supposed to be independent from AML, that would contraindicate treatment
* Subjects for which allogeneic HSCT is planned in CR1
* Known allergic or hypersensitivity to idarubicin or cytarabine or to any of the test compounds, materials
* Concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the subject at unacceptable risk
* A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 2 years
  RFS

SECONDARY OUTCOMES:
Toxicities | enitire study course until 2 years
  Number and CTC grade of all adverse events related to study treatment analyzed in an descriptive way
Minimum Residual Disease | 6, 9, 12,18 and 24 months
  Immunophenotypic characterization of human bone marrow cells will be done to determine MRD
Overall survival | 2 years
  OS

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China